CLINICAL TRIAL: NCT04054726
Title: A Study on Cerebello-Spinal tPCS in Ataxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113969
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cerebellar Ataxia
Keywords: Cerebellar ataxia; Non-invasive stimulation; Transcranial pulsed current stimulation
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tPCS (Experimental): Patients of degenerative ataxia will be randomly allocated into both the arms. Real tPCS arm will receive active tPCS. Then they will be crossed over to Sham tPCS arm.
  Interventions: Device: Active Transcranial pulsed current stimulation (tPCS)
- Sham tPCS (Sham Comparator): Patients of degenerative ataxia will be randomly allocated into both the arms. Sham tPCS arm will receive sham tPCS. Then they will be crossed over to Real tPCS arm.
  Interventions: Device: Sham Transcranial pulsed current stimulation (tPCS)

INTERVENTIONS:
Device: Active Transcranial pulsed current stimulation (tPCS) — Active tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anode will be placed on the scalp over the cerebellum area (2 cm under the inion). Cathode will be placed over the dorsal cord. Stimulation will be given for 20 mins.
  Arms: Real tPCS
Device: Sham Transcranial pulsed current stimulation (tPCS) — Sham tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anode will be placed on the scalp over the cerebellum area (2 cm under the inion). Cathode will be placed over the dorsal cord. The electric current will be ramped down 5 seconds after the beginning of the stimulation to make this condition indistinguishable from the experimental active stimulation.
  Arms: Sham tPCS

SUMMARY:
Neurodegenerative ataxia represents a group of disabling diseases. No effective treatment is currently available for them. Currently, studies are going on the effectiveness of noninvasive neurostimulation in neurodegenerative diseases. Transcranial pulsed current stimulation (tPCS) is a new modality of noninvasive neurostimulation. The investigators have planned to study the efficacy of tPCS in these patients of neurodegenerative ataxia.

Patients will be first examined clinically along with the rating of ataxia, assessment of upper limb coordination and speech as per protocol. Quantitative Electroencephalography (qEEG) and gait analysis will be done as per protocol. Next, a single session of 20 min non-invasive stimulation will be given via tPCS or sham stimulation. Stimulation will be given to cerebellum and dorsal spinal cord. After 20 mins of stimulation, re-assessment will be done using the same tools mentioned pre-stimulation.

DETAILED DESCRIPTION:
The investigators have planned to study the efficacy of cerebello-spinal stimulation via Transcranial pulsed current stimulation (tPCS) in patients of neurodegenerative ataxia. Anodal stimulation will be used for the cerebellum and cathodal stimulation for the dorsal cord.

Patients will be assessed clinically and by EEG, KinArm and Gait - before and after a single session of 20 min stimulation via tPCS or sham stimulation.

The investigators have planned to assess-

1. Speech
2. Upper limb ataxia via KinArm. Standard KinArm testing protocol will be used which is used universally.
3. Gait via Gait Carpet
4. EEG
5. Scale for the assessment and rating of ataxia (SARA)

tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anode will be placed on the scalp over the cerebellum area (2 cm under the inion). Cathode will be placed over the dorsal cord. Stimulation will be given for 20 mins.

Participant's speech will be recorded using a head-mounted microphone (AKG-c520) and a digital recording device (Zoom H4nPro) while performing the following calibrated tasks (Calibration involves a sound level meter placed at 15cm from the mouth while talker says 'ah' at 70dBA) -

1. Prolonged 'ah'.
2. Rapid repetitions of the sounds "puh", "tuh", and "kuh".
3. Two productions of a sentence with selected speech sounds (s, sh, p, b, t, i, a, u, ae, ai). "She saw Patty buy two poppies."
4. Two times louder production of a sentence with selected speech sounds. "She saw Patty buy two poppies."
5. Repetition of a continuous vowel at normal and fast rates. 'eye-eye-eye-eye-eye' without making any voice breaks or pauses".
6. Read aloud a section of a standard passage - standard rainbow passage
7. Monologue. Talk for two minutes about an interesting vacation (or an interesting hobby or activity).

The Zeno walkway will be used in conjunction with the ProtoKinetics Movement Analysis Software (PKMAS) . The walkway contains a series of pressure sensors to detect footfalls. These data will be captured and collated via the PKMAS software, resulting in numerous spatial, temporal and pressure-related gait parameters. Timed-up-and-go (TUG) task will be used, consisting of rising from chair, walking across the 20-foot gait carpet, turning around off the carpet, walking back and sitting down. This will be performed over 3 trials.

Gait analysis provides various parameters as output such as stride length, line of progression, step length, toe-offs and other temporal and spatial parameters for analysis.

Neurophysiological EEG signals will be recorded, eyes-closed, no-task, using g.Nautilus g.tec wireless system. The g.tech system uses earclip reference sensors. The subject will be in a quiet place with less light or electromagnetic perturbations. During the resting state recordings, patients are seated in a comfortable arm chair and will be instructed to keep relaxed, with their eyes closed for 5 min.

A paired t test will be used to compare baseline data and post tPCS data. Descriptive analysis of the neurological examination findings will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as neurodegenerative ataxia clinically or by genetic study.

Exclusion Criteria:

* Patients who can't walk even with support, like wheel chair bound patients.
* Patients having other issues like stroke that can aggravate speech/ gait.
* Patients who are not able to provide informed consent.
* Patients who are unable to communicate by speech and who can't comprehend the English language.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in Ataxia rating scale | 3 months
  We will evaluate the effectiveness of tPCS in patients of neurodegenerative ataxia. We will apply Scale for the assessment and rating of ataxia (SARA) for rating of ataxia pre and post stimulation. The scale is for assessing severity of ataxia, that consists of assessment of gait, stance, sitting, speech, finger chase, finger to nose test, fast alternating hand movement, heel-shin test. By summing up, the total score ranges from minimum 0 and maximum 36. Higher score means more severity.
Changes in spatiotemporal gait measures using objective gait analysis | 3 months
  We will use Zeno Walkway Gait carpet and the spatiotemporal details of the gait will be analyzed by ProtoKinetics Movement Analysis Software (PKMAS) software, pre and post stimulation.
Change in upper limb co-ordination | 3 months
  We will use KinArm pre and post stimulation to have objective measurement of upper limb co-ordination.
Change in speech | 3 months
  We will use standardized speech protocol pre and post stimulation to assess speech.
Changes in Network fragmentation using Quantitative EEG | 3 months
  We will do network fragmentation by 5 mins of resting quantitative Electroencephalography (EEG), pre and post stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258
- [Background] Alon G, Yungher DA, Shulman LM, Rogers MW. Safety and immediate effect of noninvasive transcranial pulsed current stimulation on gait and balance in Parkinson disease. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1089-95. doi: 10.1177/1545968312448233. Epub 2012 May 10. PMID 22581566
- [Background] Grimaldi G, Manto M. Anodal transcranial direct current stimulation (tDCS) decreases the amplitudes of long-latency stretch reflexes in cerebellar ataxia. Ann Biomed Eng. 2013 Nov;41(11):2437-47. doi: 10.1007/s10439-013-0846-y. Epub 2013 Jun 19. PMID 23780473
- [Background] Maas RPPWM, Toni I, Doorduin J, Klockgether T, Schutter DJLG, van de Warrenburg BPC. Cerebellar transcranial direct current stimulation in spinocerebellar ataxia type 3 (SCA3-tDCS): rationale and protocol of a randomized, double-blind, sham-controlled study. BMC Neurol. 2019 Jul 4;19(1):149. doi: 10.1186/s12883-019-1379-2. PMID 31272408